CLINICAL TRIAL: NCT05522426
Title: Open Label, Multi-Center Study, Evaluating the Effect of Adipose Tissue Processed With the SyntrFuge™ System for Facial Fat Grafting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syntr Health Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHT-SYN-02
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Facial Atrophy and Loss of Contour
Keywords: Microsized Fat Tissue; Adipose Tissue; Facial Contouring; Fat Transfer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SyntrFuge System (Experimental): Adipose tissue microsized via the SyntrFuge System
  Interventions: Device: SyntrFuge System

INTERVENTIONS:
Device: SyntrFuge System — Microsized Adipose Tissue

SUMMARY:
This is an open label multi-center study with the aim of evaluating the efficacy of adipose tissue processed with the SyntrFuge™ system in facial aesthetics and contouring. Patients will be enrolled to the treatment group with adipose tissue processed with the SyntrFuge™ system followed by an injection of autologous microsized adipose tissue in the treatment sites.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged of 18-70 years old
2. Willing and able to read and sign the informed consent and other study materials
3. Written informed consent has been obtained prior to any study-related procedures
4. Subjects are ambulatory
5. Ability to follow study instructions and complete study assessment tools including the subject diary
6. Females of childbearing potential must have a negative urine pregnancy test result and not be lactating
7. Agree to not undergo other treatments or cosmetic procedures in the treatment area during the study such as facial laser treatments, botulinum toxin, hyaluronic acid injections, any other permanent or semi-permanent facial fillers

1.5.2 Exclusion Criteria:

1. Subjects without decisional capacity
2. Subjects unable to give informed, written consent
3. Subjects with active infection (redness, swelling, pain, suppuration)
4. Subjects with any uncontrolled systemic disease
5. Subjects with a history of severe allergic/anaphylactic reactions or multiple allergies
6. Subjects with conditions within the treatment area including acne, scarring, acute lupus erythematosus, dermatitis, or melasma
7. Subjects planning to become pregnant, are pregnant, or are breast-feeding
8. Subjects with history or current evidence of drug or alcohol abuse within 12 months prior to screening visit
9. Subjects who have undergone temporary facial dermal filler injections with hyaluronic acid-based fillers within 12 months in the treatment area. Have had neuromodulator injections, mesotherapy, or resurfacing (laser or other ablative or non-ablative procedures) within 5 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study.
10. Subjects who have undergone facial plastic surgery (except for rhinoplasty or a brow lift), tissue grafting, or tissue augmentation with silicone, fat, or other permanent or semi-permanent dermal fillers or be planning to undergo any of these procedures affecting the treatment area, at any time during the study that may interfere with the study procedure and results
11. Subjects who have active autoimmune disease
12. Subjects who are unwilling to undergo fat graft injections
13. Subjects with current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
14. Subjects who have received anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti- inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen), or other substances known to increase coagulation time from 10 days pre- to 3 days post injection. A wash out period of 10 days is allowed
15. Subjects who have undergone immunosuppressive therapy, chemotherapy, biologics or systemic corticosteroids within 3 months prior to each study visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
FaceQ Satisfaction surveys | 6 months
  Change from baseline in FACE-Q Satisfaction with questionnaire score for the treated regions

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | 6 months
  Change in facial regions characteristics as measured by the Global Aesthetic Improvement Scale (GAIS) form from baseline
Investigator's Satisfaction Scale | 6 months
  Change in facial regions characteristics as measured by the Investigator's Satisfaction Scale form from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Newport Beach Site 1, Newport, California
  - Newport Beach Site 2, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No